CLINICAL TRIAL: NCT02195206
Title: DEVELOPMENT OF HYPERPOLARIZED XENON-129 LUNG AND/OR BRAIN MAGNETIC RESONANCE IMAGING HARDWARE AND SOFTWARE: HEALTHY ADULT VOLUNTEER PILOT STUDY
Brief Title: Hyperpolarized Xenon-129 Lung and/or Brain Magnetic Resonance Imaging: Healthy Adult Volunteer Pilot Study
Status: Terminated | Type: Observational
Why Stopped: Funding constraints
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Giles Santyr, PhD, FCCPM, Senior Scientist, The Hospital for Sick Children, The Hospital for Sick Children
Other Study IDs: 1000041669
Record Dates: First submitted 2014-06-19; First posted 2014-07-21 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Hyperpolarized gas magnetic resonance imaging; Hyperpolarized Xenon-129 magnetic resonance imaging; Lung and/or brain Imaging; Healthy Adults

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy: Adult

SUMMARY:
In this pilot study, MRI of the lungs and/or brain of healthy adult volunteers will be performed at 3Tesla to assess image quality using a prototype chest coil and pulse sequence following inhalation of hyperpolarized 129Xe (xenon) gas. This study will take place at the Hospital for Sick Children, Toronto, Canada. Ninety subjects aged 18 to 75 will participate in this study. Xenon MRI is a non-invasive imaging technique that does not involve X-rays or ionizing radiation. Rather, this imaging method utilizes the same hardware and software principles that are used for conventional proton MRI of patients in a hospital. The investigators are testing the abilities of xenon MRI to see if it will produce lung and/or brain images of equal or better quality to that of proton MRI.

The investigators hypothesize that they will get good quality images of the lungs and/or brain for analysis using our method.

DETAILED DESCRIPTION:
With the emergence of novel hardware and software image acquisition improvements, magnetic resonance imaging (MRI) has the potential to become an important tool for assessing lung structure and function. In particular, the use of a hyperpolarized noble gas such as 129Xe has been used to explore structural and functional relationships in the lungs of both healthy subjects and patients with lung disease (1,2). In contrast to proton-based MRI imaging, 129Xe gas is used as a "contrast agent" to directly visualize the airways, and thus image ventilation. Whereas the normal density of gas is too low to produce an easily detectable signal, this is overcome by artificially increasing the amount of polarization per unit volume using optical pumping (3).

Hyperpolarized noble gas MR lung imaging is a relatively new imaging method that allows depiction of both lung function and morphology [4-9]. Hyperpolarized gases are a new class of MR contrast agent which, when inhaled, provide high temporal and spatial resolution MR images of the lung airspaces. Since no ionizing radiation is involved, hyperpolarized gas MR imaging is ideal for the evaluation of lung diseases. With hyperpolarized gases, the nuclear spins of the gas atoms are brought into alignment outside of the MR scanner via a process called optical pumping; this yields high polarizations and permits visualization of the lung airspaces with MR imaging (despite the low physical density of the gas in the lung). Two non-radioactive (i.e. stable) isotopes of noble gases 3He and 129Xe can be hyperpolarized. Until recently, higher polarizations could be achieved with 3He than with 129Xe, so in humans, 3He was more commonly used for hyperpolarized gas MR imaging of the lungs [10-15]. Recently, the technology has been developed to provide large quantities of highly polarized 129Xe [16].

Several applications of 129Xe MRI imaging are under development, including diffusion-weighted and relaxation-weighted imaging (17-19). These techniques take advantage of the fact that the rate of loss of 129Xe polarization is significantly influenced by the local blood flow and concentration of molecular oxygen, as well as the restriction of 129Xe diffusion by small airway space dimensions. These data can be used to create maps of the lung reflecting regional ventilation/perfusion and micro-airway sizes. Other data that can be obtained with 129Xe MRI include the volumes of ventilated and unventilated lungs which can subsequently be analyzed to determine the homogeneity of gas distribution within the airspaces (17).

Another emergent application of 129Xe exploits the solubility of xenon in biological tissues and blood. This allows for the detection of 129Xe signals from beyond the airspaces, in the parenchymal lung tissue and red blood cells of the pulmonary vasculature. This enables the direct imaging and quantification of gas exchange capability of the lungs. Furthermore, xenon dissolved in the blood is carried away from the lungs to distal organs by the cardiovascular system (e.g., heart, kidneys). One organ that has seen a recent intensification of research with 129Xe is in the brain. HP 129Xe MRI of the brain holds promise for the evaluation of brain perfusion and function (31-33). Xenon dissolved in brain tissues exhibits a rich chemical shift spectrum allowing for the detection of signal from various biochemical compartments such as RBCs, cerebrospinal fluid, and white/gray matter, among others. Additionally, HP 129Xe can passively transit the blood-brain barrier in a manner that is not possible with other exogenous tracers (e.g., gadolinium-based contrast). Preliminary clinical investigations have demonstrated novelty in stroke, Alzheimer's disease, and functional brain imaging (31-33).

Objectives of the study are:

To quantitatively evaluate a 3T 129Xe radiofrequency coils (lung and/or brain) for image quality and coil comfort/performance.

To prototype and determine the range of possible novel lung and brain pulse sequences in combination with the coil and inhalation of 129Xe gas in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects male and female aged 18-75
* Subject has a smoking history of ≤ 1 pack year
* Subject understands the study procedures and is willing to participate in the study as indicated by signature on the informed consent
* Subject must be able to perform a breath hold for 16 seconds
* Subject has a Body Mass Index (BMI) between 18 and 40
* Subject is judged to be in stable health on the basis of medical history
* Subject able to perform reproducible pulmonary function tests (i.e., the 3 best acceptable spirograms have Forced Expiratory Volume (FEV1) values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater)

Exclusion Criteria:

* Subject is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material
* Subject has a history of chronic or acute respiratory disease
* Subject has a history of cardiovascular disorders including coronary insufficiency, cardiac arrhythmias, severe hypertension (≥160 over ≥100)
* Subject has a daytime room air oxygen saturation ≤ 92% ± 2% while supine
* Subject is unable to perform spirometry or plethysmography maneuvers
* Subject is pregnant or lactating
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia
* Subject has an MRI incompatible device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Adults from the general population
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Ventilation Defect Volume | Day 1
  Volume of the lung not being ventilated to the optimum level

SECONDARY OUTCOMES:
Apparent Diffusion Coefficient | Day 1
  Used to obtain structural information of the lung. Metric for assessing tissue damage.
129 Xe Brain MRI feasibility | Day 1
  129Xe brain MRI is feasible and yields images of good quality in healthy subjects.

OTHER OUTCOMES:
Signal to Noise Ratio | Day 1
  Used to assess image quality

CONTACTS AND LOCATIONS:
Overall Officials: Giles Santyr, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada